CLINICAL TRIAL: NCT00062621
Title: Combined HLA-matched Bone Marrow and Kidney Transplantation for Multiple Myeloma With Renal Failure
Brief Title: Combined Bone Marrow and Kidney Transplant for Multiple Myeloma With Kidney Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN008ST; NKDO1; DAIT NKDO1
Record Dates: First submitted 2003-06-09; First posted 2003-06-12 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Kidney Failure, Chronic; Multiple Myeloma
Keywords: Immune tolerance; Graft vs host disease; Kidney Failure; Kidney diseases; End Stage Renal Disease; Multiple Myeloma; Bone Marrow Transplant; Kidney Transplant; Renal Transplant; Tolerance; Chimerism; ESRD
MeSH Terms: conditions — Kidney Failure, Chronic; Multiple Myeloma; Graft vs Host Disease; Renal Insufficiency; Kidney Diseases | interventions — Kidney Transplantation

INTERVENTIONS:
Procedure: Combined bone marrow and kidney transplant

SUMMARY:
The purpose of this study is to determine whether a combined bone marrow and kidney transplant will be effective in treating stage II or greater multiple myeloma and associated kidney failure. This study will determine whether transplant rejection and the need for immunosuppressive drugs are decreased with this combined transplant approach.

DETAILED DESCRIPTION:
In very limited human testing, a combined kidney and bone marrow transplant appears to be safe and effective in treating multiple myeloma and associated kidney failure. This study will evaluate this approach in 10 patients with kidney failure due to or in association with stage II or greater multiple myeloma. Treatment prior to transplant will include cyclophosphamide, ATGAM (a lymphocyte-specific immunosuppressant), local radiation to the thymus, and cyclosporine (an immunosuppressive drug).

An infusion of donor bone marrow and a kidney graft from a closely matched, related donor will be transplanted simultaneously. An additional infusion of donor white blood cells may be administered between day 45 and 74 after transplant in an effort to eliminate any remaining cancer cells. Patients will remain on cyclosporine for a defined period of time. The cyclosporine doses will be slowly decreased and stopped if graft rejection and graft-versus-host disease do not occur.

Each participant will be involved in the study for 3 years; this includes the intervention phase (time from initial screening at approximately 7 days before transplant through 100 days after the transplant) and continued follow-up visits for at least 2 years following the transplant.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease (ESRD) due to or in association with stage II or greater multiple myeloma
* Participants in whom the development of ESRD is not due to the underlying myeloma will be included if they have evidence of active myeloma despite past treatment with standard therapies (e.g., prednisone, melphalan, high-dose radiation therapy with autologous stem cell transplantation)
* On dialysis or have a creatinine clearance greater than 20 ml/min
* HLA-matched or one of six HLA antigen-mismatched related donor

Exclusion Criteria:

* Compromised pulmonary, cardiac, or liver function
* Active infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2003-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Remission status of multiple myeloma | Throughout study
Renal allograft acceptance and ability to discontinue immunosuppressive therapy | Throughout study

SECONDARY OUTCOMES:
Graft vs. host disease (GVHD) | Throughout study
Opportunistic infections | Throughouto study
T-cell recovery and immune reconstitution | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spitzer, MD, Principal Investigator — Massachussetts General Hospital; A. Benedict Cosimi, MD, Principal Investigator — Massachussetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Click here for the Immune Tolerance Network Web site — http://www.immunetolerance.org
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/Pages/default.aspx